CLINICAL TRIAL: NCT03732833
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of MT10109L (NivobotulinumtoxinA) for the Treatment of Lateral Canthal Lines With or Without Concurrent Treatment of Glabellar Lines
Brief Title: MT10109L in the Treatment of Lateral Canthal Lines With or Without Concurrent Treatment of Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT10109L-006; 2014-005302-38 (EudraCT Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lateral Canthal Lines; Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- MT10109L Dose 1 + Placebo (Experimental): MT10109L Dose 1 will be injected into the LCL and Placebo into the GL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
  Interventions: Drug: MT10109L; Drug: Placebo
- MT10109L Dose 1 + MT10109L Dose 2 (Experimental): MT10109L Dose 1 will be injected into the LCL and MT10109L Dose 2 into the GL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
  Interventions: Drug: MT10109L
- Placebo (Placebo Comparator): Placebo will be injected into the LCL and into the GL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT10109L — MT10109L will be injected into either the LCL, or both the LCL and GL.
  Other Names: NivobotulinumtoxinA
  Arms: MT10109L Dose 1 + MT10109L Dose 2; MT10109L Dose 1 + Placebo
Drug: Placebo — Placebo will be injected into either the GL, or both the LCL and GL.
  Arms: MT10109L Dose 1 + Placebo; Placebo

SUMMARY:
To evaluate the safety and efficacy of MT10109L for the treatment of lateral canthal lines (LCL) with or without concurrent treatment of glabellar lines (GL) in participants with moderate to severe LCL and GL.

ELIGIBILITY:
Inclusion Criteria:

-Female participants must not be pregnant or planning to get pregnant and willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period.

Exclusion Criteria:

* Known immunization or hypersensitivity to any botulinum toxin serotype.
* Any medical condition that may put the participant at increased risk with exposure to MT10109L including diagnosed myasthenia gravis, Eaton Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
* History of facial nerve palsy.
* Any uncontrolled systemic disease.
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study intervention).
* Anticipated need for surgery or overnight hospitalization during the study.
* Prior exposure to botulinum toxin of any serotype for any reason.
* Prior periorbital surgery, facial lift (full face or mid-face), thread lift, brow lift, or related procedures (eg, eyelid [blepharoplasty] and/or eyebrow surgery).
* Prior facial treatment with permanent soft tissue fillers, synthetic implantation (eg, Gore-Tex®), and/or autologous fat transplantation.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Females who are pregnant, nursing, or planning a pregnancy during the study.
* Participants who plan for an extended absence away from the immediate area of the study site that would preclude them from returning for all protocol-specified study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SangMi Park, Study Director — Medytox Inc
Locations (20):
- United States (11):
  - Clear Dermatology & Aesthetics Center, Scottsdale, Arizona
  - Art of Skin MD, Solana Beach, California
  - Susan H. Weinkle, MD, Bradenton, Florida
  - Etre Cosmetic Dermatology and Laser Center, New Orleans, Louisiana
  - Dermatology and Laser Surgery Center of New York, New York, New York
  - Skin Search of Rochester Inc., Rochester, New York
  - M3 Wake Research Inc., Raleigh, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Aventiv Research Inc., Dublin, Ohio
  - Westlake Dermatology & Cosmetic Surgery - Westlake, Austin, Texas
  - DermResearch Inc., Austin, Texas
- Canada (4):
  - Dr. Jean Carruthers Cosmetic Surgery Inc., Vancouver, British Columbia
  - Pacific Derm, Vancouver, British Columbia
  - Dermetics Cosmetic Dermatology, Burlington, Ontario
  - Nectar Research Group Inc., Richmond Hill, Ontario
- Germany (5):
  - Rosenpark Research, Darmstadt, Hesse
  - Hautzentrum Koln - Cologne Dermatology, Cologne
  - Hautok and Hautok-cosmetics, München
  - MediCorium Zentrum fuer Dermatologie und Aesthetik, Oberursel
  - CentroDerm GmbH, Wuppertal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 602 participants were screened, 424 participants were analyzed in ITT set and 425 participants were analyzed in Safety set.
Groups:
- Placebo: Placebo was injected into the Lateral Canthal Lines (LCL) and into the Glabellar Lines (GL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
- MT10109L 24U + Placebo: MT10109L 24U was injected into the Lateral Canthal Lines (LCL) and Placebo into the Glabellar Lines (GL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
- MT10109L 24U + MT10109L 20U: MT10109L 24U was injected into the Lateral Canthal Lines (LCL) and MT10109L 20U into the Glabellar Lines (GL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
Period: Overall Study
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Started | 86 | 171 | 167 (The number of participants in the Efficacy set = 167; The number of participants in the Safety set = 168)
Completed | 68 | 138 | 150
Not Completed | 18 | 33 | 17
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Withdrawal by Subject | 11 | 13 | 8
Not completed — Lost to Follow-up | 3 | 5 | 4
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Physician Decision | 2 | 3 | 1
Not completed — Covid-19 related and other reasons | 2 | 7 | 3

BASELINE CHARACTERISTICS:
Population: 424 participants were included in the ITT population (86 in the Placebo; 171 in the MT10109L 24 U group and 167 participants in the MT10109L 44U group)
Groups:
- MT10109L 24U + Placebo: MT10109L 24U was injected into the Lateral Canthal Lines (LCL) and Placebo into the Glabellar Lines (GL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
  .
- Total: Total of all reporting groups
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U | Total
Number analyzed (Participants) | 86 | 171 | 167 | 424
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 156 | 157 | 393
  >=65 years | 6 | 15 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.32) | 47.7 (11.56) | 49.1 (10.37) | 48.5 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 143 | 141 | 355
  Male | 15 | 28 | 26 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 10 | 25
  Not Hispanic or Latino | 82 | 159 | 157 | 398
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 0 | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 3 | 8
  White | 85 | 161 | 159 | 405
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the Facial Wrinkle Scale With Photonumeric Guide (FWS) According to INVESTIGATOR AND PARTICIPANT Assessments of LCL Severity at Maximum Smile at Day 30
Description: The outcome measured is the percentage of participants who had a ≥2-grade improvement from baseline LCL severity at maximum smile according to investigator and participant FWS ratings at Day 30.
  Both the INVESTIGATOR AND PARTICIPANT evaluate the LCL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe. The primary endpoint is achieved and recorded as a count only when BOTH INVESTIGATOR AND PARTICIPANT assess the improvement in FWS from baseline to be ≥ 2-grade improvement. Therefore, the primary endpoint is the proportion/percentage of participants who meet the dual assessment threshold of ≥2-grade improvement from baseline.
Time Frame: Day 30
Population: The primary endpoint measurements were carried out using the Intent-To-Treat (ITT) analysis set, which was defined as all participants who were randomized. Multiple imputation method was used for missing variables in primary efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 86 | 171 | 167
Participants | 0 | 35 | 38

2. Secondary Outcome: The Percentage of Responders for INVESTIGATOR Assessments of Lateral Canthal Lines (LCL) Severity at Maximum Smile Using the Facial Wrinkle Scale With Photonumeric Guide (FWS)
Description: The outcome here only considers the INVESTIGATOR assessments (excludes the participant assessment). The investigator evaluates the participant's LCL severity using a 4-point scale (0 to 3) where 0=none and 3=severe. A Responder was defined as one achieving a ≥2-grade improvement from baseline at maximum smile at Day 30.
Time Frame: Day 30
Population: All secondary efficacy analyses were carried out using the Intent-To-Treat (ITT) analysis subset, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo was injected into the Lateral Canthal Lines (LCL) and into the Glabellar Line (GL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 80 | 164 | 166
Participants | 0 | 59 | 64

3. Secondary Outcome: The Duration of Lateral Canthal Lines (LCL) Treatment in Participants Who Achieved a Rating of ≥ 2-grade Improvement From Baseline in LCL Severity at Maximum Smile at Day 30 According to Investigator Assessments Using the FWS
Description: The investigator evaluates the participant's LCL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Time Frame: Day 1 (first treatment) to Day 180
Population: All secondary efficacy analyses were carried out using the Intent-To-Treat (ITT) analysis subset, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data. The participant analyzed here corresponds to the responders in Outcome 2.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Placebo: Placebo was injected into the LCL and into the GL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
- MT10109L 24U + Placebo: MT10109L 24U was injected into the LCL and Placebo into the GL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
- MT10109L 24U + MT10109L 20U: MT10109L 24U was injected into the LCL and MT10109L 20U into the GL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 0 | 59 | 64
Days |  | 113 [91 to 121] | 93 [89 to 118]

4. Secondary Outcome: The Percentage of Participants Reporting Mostly Satisfied/Very Satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 for Lateral Canthal Lines (LCL)
Description: The Satisfaction Question 5 grades facial line treatment satisfaction on a 5-point scale (-2 to 2) where -2=Very dissatisfied and 2=Very satisfied.
Time Frame: Day 60
Population: All secondary efficacy analyses were carried out using the Intent-To-Treat (ITT) analysis set or subset, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 75 | 158 | 156
Participants | 8 | 97 | 122

5. Secondary Outcome: The Percentage of Responders for Investigator Assessments of Lateral Canthal Lines (LCL) Severity at Rest Using the Facial Wrinkle Scale (FWS)
Description: The investigator evaluates the participant's LCL severity using a 4-point scale (0 to 3) where 0=none and 3=severe.
  Among Participants Who Were Rated At least Mild at Rest at Baseline, where a Responder was Defined as Achieving a ≥1-grade Improvement from Baseline at Day 30. The outcome measured here is the proportion of participants who achieved a ≥1-grade improvement from baseline LCL severity at rest based on investigator FWS rating.
Time Frame: Day 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 77 | 158 | 158
Participants | 13 | 106 | 107

6. Secondary Outcome: Number of Patients Who Experienced a Treatment Emergent Adverse Event (TEAEs)
Description: This section focuses primarily on TEAEs, i.e., AEs that started or worsened after the first dose of study intervention and within 30 days after the last dose. The safety analyses were conducted in the Safety population. Unless otherwise noted, safety results refer to TEAEs.
Time Frame: AEs that started or worsen after the first dose of study intervention and within 30 days after the last dose.
Population: All safety analyses were carried out using the Safety population set or subset, defined as participants who received at least 1 dose of study intervention. Participants were grouped based on their actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 86 | 171 | 168
Participants | 50 | 90 | 106

7. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (BP)
Description: The outcome reported here is the mean change in Systolic BP from baseline to study exit.
Time Frame: Baseline to Day 360
Population: The population analyzed for this outcome was the subset of participants from the Safety population remaining at study exit. Participants were grouped based on their actual treatment received.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 73 | 149 | 157
mmHg | 1.0 (11.60) | -0.4 (12.29) | -0.3 (13.67)

8. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (BP)
Description: The outcome reported here is the mean change in Diastolic BP from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 73 | 149 | 157
mmHg | -1.2 (8.61) | -1.4 (8.34) | -0.7 (9.28)

9. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Description: The outcome reported here is the mean change in Pulse Rate from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 73 | 149 | 157
beats/min | -0.7 (11.2) | 0.9 (10.54) | -0.4 (11.34)

10. Secondary Outcome: Mean Change From Baseline in Respiratory Rate
Description: The outcome reported here is the mean change in Respiratory Rate from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 73 | 149 | 157
breaths/min | -0.4 (2.03) | -0.3 (2.04) | -0.6 (2.47)

11. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - Mean Heart Rate
Description: The outcome reported here is a mean change in mean heart rate from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 72 | 149 | 157
beats/min | 3.3 (10.34) | 4.2 (9.35) | 2.7 (8.34)

12. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - PR Interval
Description: The outcome reported here is a mean change in PR interval from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 71 | 149 | 157
milliseconds | -0.5 (9.36) | -0.7 (12.37) | 0.0 (11.09)

13. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QRS Duration
Description: The outcome reported here is a mean change in QRS duration from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 72 | 149 | 157
milliseconds | 0.0 (6.16) | 0.4 (5.35) | 1.6 (8.06)

14. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QT Interval
Description: The outcome reported here is a mean change in QT interval from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 72 | 149 | 157
milliseconds | -8.6 (25.07) | -10.4 (21.96) | -9.2 (21.26)

15. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcB Interval
Description: The outcome reported here is a mean change in QTcB interval from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 72 | 149 | 157
milliseconds | 0.9 (17.34) | 1.6 (16.64) | -1.5 (16.3)

16. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcF Interval
Description: The outcome reported here is a mean change in QTcF interval from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 72 | 149 | 157
milliseconds | -2.4 (14.21) | -2.7 (13.57) | -4.2 (13.65)

17. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - RR Interval
Description: The outcome reported here is a mean change in RR interval from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 72 | 149 | 157
milliseconds | -42.6 (137.27) | -53.0 (120.85) | -35.0 (114.66)

18. Secondary Outcome: Number of Participants With Binding and Neutralizing Antibodies
Description: Only samples that tested positive in the binding antibody confirmatory assay were evaluated for neutralizing antibodies. The participants with positive neutralizing antibodies are only shown.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
Number analyzed (Participants) | 72 | 145 | 150
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: This section describes Treatment-Emergent Adverse Events (TEAEs) that started or worsened after the first dose of study intervention and within 30 days after the last visit or study exit (Day 360 unless the participant exits earlier)
Description: Treatment-emergent adverse events were classified according to MedDRA, Version 23.1.
Arm/Group | Placebo | MT10109L 24U + Placebo | MT10109L 24U + MT10109L 20U
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/171 | 0/168
Serious Adverse Events (participants affected / at risk) | 4/86 | 11/171 | 5/168
Other Adverse Events (participants affected / at risk) | 34/86 | 60/171 | 74/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=86) | MT10109L 24U + Placebo (N=171) | MT10109L 24U + MT10109L 20U (N=168)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 2 (2)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion induced [F] (Surgical and medical procedures) | 0/71 (0) | 1/143 (1) | 0/141 (0) — Calculated with respect to number of Female participants at risk
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=86) | MT10109L 24U + Placebo (N=171) | MT10109L 24U + MT10109L 20U (N=168)
Headache (Nervous system disorders) | 3 (3) | 9 (9) | 22 (22)
Nasopharyngitis (Infections and infestations) | 6 (6) | 16 (16) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4) | 10 (10)
Injection site pain (General disorders) | 8 (8) | 15 (15) | 15 (15)
Injection site haemorrhage (General disorders) | 6 (6) | 9 (9) | 6 (6)
Injection site bruising (General disorders) | 6 (6) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
General research agreement between the sponsor and PI's that includes a confidentiality section that includes a statement that the sponsor is and shall remain the exclusive owner of 'Information'. ) 'Information' shall include, but shall not be limited to, protocols, trade secrets, know-how, formulations, inventions, techniques, equipment, data and results.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03732833/Prot_004.pdf
  • Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03732833/SAP_006.pdf